CLINICAL TRIAL: NCT07041268
Title: Evaluation of Effectiveness and Safety of the Rituximab Immunotherapy Plus Insulin Therapy Compared to Insulin Therapy Alone in Adolescents With Recent-Onset Type 1 Diabetes Mellitus
Brief Title: Immunotherapy of the Recent-onset Type 1 Diabetes in Adolescents With Repeated Courses of Rituximab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-11-14
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Rituximab

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Rituximab Plus Insulin Therapy Arm (Experimental): In the Rituximab Plus Insulin Therapy Arm, patients will receive repeated courses of rituximab along with their routine insulin therapy
  Interventions: Biological: rituximab
- Insulin Therapy Only Arm (No Intervention): In the Insulin Therapy Only Arm, patients will receive their routine insulin therapy

INTERVENTIONS:
Biological: rituximab — Rituximab will be administered intravenously in three courses. The 1st course (loading dose) will include six rituximab infusions on days 1, 3, 5, 8, 14, and 21 of the study. On days 1, 3, and 5 rituximab will be infused at doses of 50, 125, and 200 mg per m2 of the participant's body surface area, respectively. On days 8, 14, and 21 rituximab will be infused at doses of 375 mg/m2, but not more than 500 mg total dose.
  The 2nd course (maintenance therapy) will include four rituximab infusions on days 63, 70, 77, and 85 at doses of 375 mg/m2, but not more than 500 mg total dose.
  The 3rd course (maintenance therapy) will include four rituximab infusions on days 119, 126, 134, and 140 at doses of 375 mg/m2, but not more than 500 mg total dose
  Arms: Intervention Arm: Rituximab Plus Insulin Therapy Arm

SUMMARY:
Type 1 diabetes (T1D) is caused by destruction of pancreatic islet beta-cells that produce insulin - the hormone required for glucose uptake by body tissues and organs. Since loss of beta-cells leads to insulin deficiency, blood glucose increases and the symptoms of T1D (thirst, hunger, excessive urination) appear. Inability of patient's tissues and organs to utilize glucose results in rapid weight loss and life-threatening acute T1D complications - ketosis and coma. To ensure glucose consumption by tissues and organs and to prevent acute complications, all patients with T1D need lifelong therapy with insulin. Insulin therapy is also necessary to prevent long-term T1D complications (eye, renal, nerve, and heart problems). By the time T1D is diagnosed, 80-90% of beta-cells have already been destroyed. However, 10-20% viable insulin-producing beta-cells remain in the pancreas over several months and even years after T1D diagnosis. The higher the percentage of the remaining beta-cells, the smaller the risk of long-term complications.

Destruction of beta-cells in T1D has an autoimmune origin. It means that the patient's immune system, which is normally targeted at microbes, viruses, and other non-self substances, mistakenly destroys the beta-cells. The key role in this autoimmune reaction is played by specific cells of the immune system: T- and B-lymphocytes. T-lymphocytes directly damage the beta-cells, while B-lymphocytes support T-lymphocytes activity via antigen presentation mechanisms.

Rituximab is a drug that specifically eliminates B-lymphocytes from the blood based on the CD20 surface molecule expressed on their surface, as a target. Notably, a subset of currently active T cells, including those potentially associated with pathogenesis of multiple sclerosis, also express CD20 marker on their surface. This makes them a potentially another critically important target of rituximab. In 2009 - 2014, a multicenter study in the U. S. and Canada showed that a single three-week course of rituximab infusions slightly but significantly had improved survival of residual beta-cells and their insulin-producing capacity in patients with recent-onset T1D. However, this beneficial action of rituximab lasted for only one year.

We hypothesized that the repeated courses of rituximab performed over a period of 5 months could produce more profound and durable elimination of pathogenic B- and T- cells, and as a consequence prolonged survival of residual beta-cells and insulin secretion without serious adverse events. Testing this hypothesis is the goal of our study

DETAILED DESCRIPTION:
The study is a non-randomized, two-arm, open-label trial in which 1/2 of participants will receive repeated infusions of rituximab and their routine insulin therapy, while the remaining 1/2 will receive their routine insulin therapy only). The group the participant is assigned to is chosen by the participant himself/herself, participant's parent or another legally authorized representative, and by a doctor at the study Clinical Center. In the rituximab group, participants will receive fourteen intravenous infusions of rituximab over a period of 1 year at the study Clinical Center. Over this period, the participants will need to return to the Clinical Center for hospitalization 13 times. At each visit, detailed physical examination and laboratory evaluation will be performed. Participants of the insulin-only group will also need to visit the Clinical Center for physical examination and laboratory evaluation 5 times over a period of 1 year. In both groups, beta-cell survival and insulin-secreting capacity will be assessed by measuring blood C-peptide levels. C-peptide is a small protein secreted by beta-cells together with insulin in equal amounts, thus allowing to assess beta-cell secretory activity in individuals receiving insulin therapy. C-peptide will be measured in the fasting state and at 15, 30, 60, 90, and 120 minutes after oral liquid meal load. This test will be performed at the study start and in the 12th, 19th, 26th, and 52nd week after the start.

In both groups, those participants that continue to secrete insulin will have further follow-up for an additional one year

ELIGIBILITY:
Inclusion Criteria:

* Is 12 years to 17 years 5 months of age, inclusive, at the time of randomization/initiation of rituximab administration
* Body weight 34-80 kg for males, and 37-80 for females
* Has received a diagnosis of type 1 diabetes mellitus (T1D), ICD-10 codes E10.1 or E10.9, according to the criteria from the Russian Association of Endocrinologists
* The duration of T1D (time from diagnosis to screening) is < 4 months
* Is able to be randomized and initiate rituximab infusions within 4 months (122 days) of the formal T1D diagnosis
* Has a peak stimulated C-peptide of ≥ 200 pmol/L from a MMTT at screening
* Is positive for at least one of T1D-related autoantibodies (ICA, GADA, IA-2A, ZnT8A) at screening
* Participant AND his/her legally authorized representative have signed the Informed Consent Form
* Citizenship of the Russian Federation

Exclusion Criteria:

* Has any autoimmune disease other than T1D with the exception of stable thyroid or celiac disease
* Has an active infection and/or fever
* Has a history of or serologic evidence of current or past infection with Mycobacterium tuberculosis, human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at screening
* Has a history of primary immunodeficiency
* Has a medical, psychological or social condition that, in the opinion of the Principal Investigator, would interfere with safe and proper completion of the trial
* Participant AND his/her legally authorized representative have not signed the Informed Consent Form

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Mean C-peptide Area Under Curve (AUC) Standardized by Duration of the Mixed Meal Tolerance Test | In the Rituximab Plus Insulin Therapy Arm, MMTT will be conducted on study days -1 (the day before the first rituximab infusion), 84, 133, 181, and 365. In the Insulin Therapy Only Arm, MMTT will be conducted on study days 1, 84, 133, 181, and 365
  Calculation of the AUC is based on serum C-peptide measurements performed at 0, 15, 30, 60, 90, and 120 minutes of the MMTT. The AUC is computed using the trapezoidal rule and standardized by the duration of the MMTT, i.e., the mean AUC is expressed algebraically as the AUC/120 min (picomoles/liter/120 min). Commercial nutritional drink is used as a load for MMTT. The drink volume and carbohydrate content are adjusted to participant's weight

SECONDARY OUTCOMES:
Change in Average Daily Insulin Dose | Baseline to Day 365
  The average weight-ajusted daily insulin dose will be calculated based on data recorded by participants in their electronic diary (eDiary). Will be assessed in both arms
Change in Glycosylated Hemoglobin | Baseline to Day 365
  Change in content of glycosylated hemoglobin HbA1c in blood, % and mmol/mol. Will be assessed in both arms
Time in Range for Glycemia Control | Baseline to Day 365
  Time in range (%) for glycemia control will be assessed using participant's continuous glucose monitoring (CGM) or flash glucose monitoring (FGM) device. Time in range is defined as daily average percentage of time a participant's glucose is ≥ 3.9 mmol/L and <10 mmol/L. Will be assessed in both arms
Frequency of Clinically Significant Hypoglycemia | Baseline to Day 365
  Frequency here = (clinically significant hypoglycemic episode)/(participant-year). A clinically significant hypoglycemia is defined as a blood glucose level of <3.0 mmol/L or a hypoglycemia episode with severe cognitive impairment requiring external assistance (seizure, syncope, severe confusion) with or without a confirmatory low blood glucose. Hypoglycemia frequency will be calculated for each participant as (number of episodes)/365 days. The number of hypoglycemic episodes will be extracted from participant's eDiary. Will be assessed in both arms

OTHER OUTCOMES:
Number of Participants With Adverse Events | During the entire study (from the first rituximab infusion to the last contact with the participant up to 365 days
  Will be assessed only in the Rituximab Plus Insulin Therapy Arm (intervention arm)
Anti-Rituximab Antibody (ARitA) Titers | Days 63, 70, 77, 85, 119, 126, 134, 140, 181, and 365
  ARitA in serum will be measured by ELISA in the Rituximab Plus Insulin Therapy Arm (intervention arm) only
Anti-Beta-Cell Antibody (ABCA) Titers | Days 0, 70, 85, 134, 140, 181, and 365
  ABCA will include determinations of serum autoantibodies to glutamic acid decarboxylase (GAD65), thyrosine phosphatase/Islet Antigen 2 (IA-2), zinc transporter 8 (ZnT8) by ELISA and cytoplasmic islet cell antibodies (ICA) by indirect immunofluorescence. ABCA will be measured in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry M Chudakov, Ph.D., D.Sc., Study Chair — Institute of Translational medicine, Pirogov Russian National Research Medical University; Elena E Petryaykina, M.D., Study Director — Russian Children's Clinical Hospital, Pirogov Russian National Research Medical University; Elena S Demina, M.D., Principal Investigator — Russian Children's Clinical Hospital, Pirogov Russian National Research Medical University
Locations (2):
- Russia (2):
  - I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow
  - Russian Children's Clinical Hospital, Pirogov Russian National Research Medical University, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pescovitz MD, Greenbaum CJ, Bundy B, Becker DJ, Gitelman SE, Goland R, Gottlieb PA, Marks JB, Moran A, Raskin P, Rodriguez H, Schatz DA, Wherrett DK, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet Anti-CD20 Study Group. B-lymphocyte depletion with rituximab and beta-cell function: two-year results. Diabetes Care. 2014 Feb;37(2):453-9. doi: 10.2337/dc13-0626. Epub 2013 Sep 11. PMID 24026563
- [Background] Greenbaum CJ, Mandrup-Poulsen T, McGee PF, Battelino T, Haastert B, Ludvigsson J, Pozzilli P, Lachin JM, Kolb H; Type 1 Diabetes Trial Net Research Group; European C-Peptide Trial Study Group. Mixed-meal tolerance test versus glucagon stimulation test for the assessment of beta-cell function in therapeutic trials in type 1 diabetes. Diabetes Care. 2008 Oct;31(10):1966-71. doi: 10.2337/dc07-2451. Epub 2008 Jul 15. PMID 18628574
- See also: Contains the complete version of the Study Protocol (in Russian) — https://static-0.minzdrav.gov.ru/system/attachments/attaches/000/062/176/original/2023-11-14.pdf?1686728191